CLINICAL TRIAL: NCT01624961
Title: Controlled Human Malarial Infection by Intravenous Injection of Plasmodium Falciparum Sporozoites in Non-Immune Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Institute of Tropical Medicine, University of Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TUCHMI-001
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Malaria
Keywords: Controlled human malaria infection (CHMI); Malaria challenge; Plasmodium falciparum; PfSPZ Challenge
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 50 PfSPZ IV (Experimental): PfSPZ Challenge
  Interventions: Biological: PfSPZ Challenge
- 200 PfSPZ IV (Experimental): PfSPZ Challenge
  Interventions: Biological: PfSPZ Challenge
- 800 PfSPZ IV (Experimental): PfSPZ Challenge
  Interventions: Biological: PfSPZ Challenge
- 3200 PfSPZ IV (Experimental): PfSPZ Challenge
  Interventions: Biological: PfSPZ Challenge
- 2500 PfSPZ ID (Experimental): PfSPZ Challenge
  Interventions: Biological: PfSPZ Challenge

INTERVENTIONS:
Biological: PfSPZ Challenge — PfSPZ Challenge are aseptic, cryopreserved P. falciparum sporozoites.
  Other Names: Aseptic, cryopreserved P. falciparum sporozoites

SUMMARY:
The study is designed to establish the best dose to safely infect healthy individuals with Plasmodium falciparum sporozoites (PfSPZ) via intravenous (IV) injection.

DETAILED DESCRIPTION:
TÜCHMI-001 is a single center, open label, randomized and controlled human pilot study to optimize controlled human malaria infection(CHMI) administered by PfSPZ Challenge. Volunteers will be inoculated with PfSPZ Challenge. Controls will receive the PfSPZ Challenge by ID administration. The remaining volunteers will receive the PfSPZ Challenge by IV administration. All volunteers recruited will be healthy adults aged between 18 and 45 years. Safety and infectivity data will be collected for each of the regimens and dose-levels.

Volunteers and clinical investigators will not be blinded to group allocation, however laboratory investigators processing blood films and samples for PCR analysis will be blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner if required
* Women only: Must agree to practice continuous effective contraception for the duration of the study (a method which results in a low failure rate; i.e. less than 1% per year)
* Agreement to refrain from blood donation during the course of the study and after the end of their involvement in the study according to the local blood banking eligibility criteria
* Written informed consent to undergo CHMI
* Reachable (24/7) by mobile phone during the whole study period
* Willingness to take a curative anti-malarial regimen
* Agreement to stay overnight for observation during the period of intensive follow-up post-challenge if required
* Answer all questions on the informed consent quiz correctly
* A body mass index <35
* A haemoglobin concentration ≥12 g/dl for women and ≥14 g/dl for men

Exclusion Criteria:

* History of P. falciparum malaria
* History of long term residence (>5 years) in area known to have significant transmission of P. falciparum
* Use of systemic antibiotics with known antimalarial activity within 30 days of study enrolment (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones, or azithromycin)
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period
* Prior receipt of an investigational malaria vaccine
* HIV infection
* Any confirmed or suspected immunosuppressive or immunodeficient state, asplenia, recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* Use of immunoglobulins or blood products within 3 months prior to enrolment
* Presence of sickle cell anemia, sickle cell trait, thalassemia or thalassemia trait
* Pregnancy, lactation or intention to become pregnant during the study
* A history of allergic disease or reactions likely to be exacerbated by malaria
* Contraindications to the use of the first-line anti-malarial medications: Atovaquone/Proguanil, Artemether/Lumefantrine, and Chloroquine
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition that may affect participation in the study
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 60g (men) or 40g (women) per day
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Falling in moderate risk or higher categories for fatal or non-fatal cardiovascular event within 5 years (>10%) determined by non-invasive criteria for cardiac risk
* Abnormal electrocardiogram on screening: pathologic Q wave and significant ST-T wave changes, left ventricular hypertrophy, non-sinus rhythm except isolated premature atrial contractions, right of left bundle branch block, advanced A-V heart block (secondary or tertiary)
* A QT/QTc interval >450 ms
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination
* Any other significant disease, disorder or finding which, in the opinion of the Investigator, may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The infectivity of the administration regimens will be assessed by thick film microscopy and PCR for P. falciparum DNA. | Day 5 until day 21 or until treatment
  Parasitology and parasite molecular biology tests: These tests are used to determine malaria parasites (thick blood smear and PCR). Both tests are performed at screening and then approximately every 12 hours during the period of intense observation from day 5 until day 21 or until treatment. Thereafter, these tests are performed during safety follow-ups at Days 28, 84, and 168. Turn over time for thick blood smear microscopy is < 2 hours to ensure timely treatment in case of a positive result. PCR results are available only after study completion.

SECONDARY OUTCOMES:
The time from parasite inoculation to first detection of blood stage parasitemia will be assessed by thick blood film microscopy. | Day 5 until day 21 or until treatment
The safety of PfSPZ Challenge administered ID or IV and the resultant P. falciparum infection will be assessed by analysing actively and passively collected data from clinical review of volunteers and laboratory measurements | Screening to Day 168
  These tests include full blood picture (complete blood count), liver enzymes and creatinine. All of these will be performed once at screening, Day -1 (day before challenge), Day 21 when no parasitemia occurs until then and day of malaria diagnosis. Lastly, these tests will also be performed during safety follow up at Days 28, 84 and 168.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin G Mordmüller, MD, Principal Investigator — Eberhard Karls University of Tübingen, Germany
Locations (1):
- Eberhard Karls University of Tübingen, Germany, Tübingen, Germany

REFERENCES:
- [Background] Gomez-Perez GP, Legarda A, Munoz J, Sim BK, Ballester MR, Dobano C, Moncunill G, Campo JJ, Cistero P, Jimenez A, Barrios D, Mordmuller B, Pardos J, Navarro M, Zita CJ, Nhamuave CA, Garcia-Basteiro AL, Sanz A, Aldea M, Manoj A, Gunasekera A, Billingsley PF, Aponte JJ, James ER, Guinovart C, Antonijoan RM, Kremsner PG, Hoffman SL, Alonso PL. Controlled human malaria infection by intramuscular and direct venous inoculation of cryopreserved Plasmodium falciparum sporozoites in malaria-naive volunteers: effect of injection volume and dose on infectivity rates. Malar J. 2015 Aug 7;14:306. doi: 10.1186/s12936-015-0817-x. PMID 26245196
- [Result] Mordmuller B, Supan C, Sim KL, Gomez-Perez GP, Ospina Salazar CL, Held J, Bolte S, Esen M, Tschan S, Joanny F, Lamsfus Calle C, Lohr SJ, Lalremruata A, Gunasekera A, James ER, Billingsley PF, Richman A, Chakravarty S, Legarda A, Munoz J, Antonijoan RM, Ballester MR, Hoffman SL, Alonso PL, Kremsner PG. Direct venous inoculation of Plasmodium falciparum sporozoites for controlled human malaria infection: a dose-finding trial in two centres. Malar J. 2015 Mar 18;14:117. doi: 10.1186/s12936-015-0628-0. PMID 25889522
- [Derived] Requena P, Gomez-Perez GP, McCall MBB, Barrios D, Aguilar R, Fernandez-Morata J, Vidal M, Campo JJ, Sanchez C, Yazdabankhsh M, Sim BKL, Hoffman SL, Kremsner P, Lell B, Mordmuller B, Dobano C, Moncunill G. Effect of controlled human Plasmodium falciparum infection on B cell subsets in individuals with different levels of malaria immunity. Med Microbiol Immunol. 2025 Sep 27;214(1):47. doi: 10.1007/s00430-025-00847-x. PMID 41014333
- See also: Publication of trials results — http://www.malariajournal.com/content/14/1/117